CLINICAL TRIAL: NCT05129215
Title: Development and Validation of a Nomogram to Predict Severe Bowel Dysfunction After Rectal Cancer Resection and Neoadjuvant Radiotherapy: A Multicenter, Observational Clinical Study
Brief Title: Development and Validation of The Post-RT LARS Prediction Model (PORTLARS)
Acronym: PORTLARS
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E2020016
Record Dates: First submitted 2021-11-15; First posted 2021-11-22 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Low Anterior Resection Syndrome; Radiotherapy; Rectal Cancer
Keywords: Bowel Dysfunction; Low Anterior Resection Syndrome; Radiotherapy; Rectal Cancer
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms; Intestinal Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Development: A primary cohort of eligible patients from the Sixth Affiliated Hospital of Sun Yat-sen University is used for model derivation.
  Interventions: Other: Questionnaire
- Internal cross-validation: A cohort of consecutive patients from the Sixth Affiliated Hospital of Sun Yat-sen University is used for internal cross-validation.
  Interventions: Other: Questionnaire
- External validation: An independent cohort of eligible patients from other hospitals is used for external validation.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The LARS score is used for assessment of bowel dysfunction after rectal cancer resection.

SUMMARY:
Bowel dysfunction is common after a restorative rectal cancer resection. Neoadjuvant radiotherapy is an influential factor that impairs bowel function and quality of life. However, almost half patients who have received primary surgery with preoperative radiotherapy are able to restore a good or moderate bowel function in the long term. This multicenter observational study aims to identify the risk factors of severe bowel dysfunction after rectal cancer resection and neoadjuvant radiotherapy, in accordance with the LARS score, and to build a model that predicts long-term major LARS in the early stage of follow-up. Development and validation cohorts are enrolled from tertiary hospitals in China.

ELIGIBILITY:
Inclusion Criteria:

* Curative low anterior resection for nonmetastatic rectal cancer
* Preoperative radiotherapy

Exclusion Criteria:

* Death
* Metastasis or recurrence
* Postoperative radiotherapy
* Cognitive disorder
* Intestinal stoma
* Rectal cancer resection for <12 months
* Stoma reversal for <6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent preoperative radiotherapy and curative low anterior resection for nonmetastatic rectal cancer.
Sampling Method: Probability Sample
Enrollment: 901 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) | Over one year after restorative rectal cancer resection
  The AUC of PORTLARS in predicting major bowel dysfunction after restorative rectal cancer resection with neoadjuvant radiotherapy.
  The AUC is evaluated by calculating the area under curve of receiver operating characteristics which plots the proportion of true positive cases (sensitivity) against the proportion of false positive cases (1-specificity) based on various predictive probability threshold.

SECONDARY OUTCOMES:
Sensitivity | Over one year after restorative rectal cancer resection
  The sensitivity of PORTLARS in predicting major bowel dysfunction after restorative rectal cancer resection with neoadjuvant radiotherapy.
  Model sensitivity is evaluated by calculating the proportion of the 'predicted major LARS' subjects among the total 'actual major LARS' subjects.
Specificity | Over one year after restorative rectal cancer resection
  The specificity of PORTLARS in predicting major bowel dysfunction after restorative rectal cancer resection with neoadjuvant radiotherapy.
  Model specificity is evaluated by calculating the proportion of the 'predicted no/minor LARS' subjects among the total 'actual no/minor LARS' subjects.
Positive prediction value (PPV) | Over one year after restorative rectal cancer resection
  The PPV of PORTLARS in predicting major bowel dysfunction after restorative rectal cancer resection with neoadjuvant radiotherapy.
  Model PPV is evaluated by calculating the proportion of the 'actual major LARS' subjects among the total 'predicted major LARS' subjects.
Negative prediction value (NPV) | Over one year after restorative rectal cancer resection
  The NPV of PORTLARS in predicting major bowel dysfunction after restorative rectal cancer resection with neoadjuvant radiotherapy.
  Model NPV is evaluated by calculating the proportion of the 'actual no/minor LARS' subjects among the total 'predicted no/minor LARS' subjects.

OTHER OUTCOMES:
Net reclassification index (NRI) | Over one year after restorative rectal cancer resection
  The additive NRI of PORTLARS compared to other models is evaluated by calculating the percentage of the 'actual major LARS' subjects correctly reclassified to the percentage of the 'actual no/minor LARS' subjects who are correctly reclassified.

CONTACTS AND LOCATIONS:
Overall Officials: Qiyuan Qin, M.D., Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Qin Q, Huang B, Wu A, Gao J, Liu X, Cao W, Ma T, Kuang Y, Guo J, Wu Q, Shao B, Guan Q, Yao H, Zhang X, Wang H; Chinese Radiation Intestinal Injury Research Group. Development and Validation of a Post-Radiotherapy Prediction Model for Bowel Dysfunction After Rectal Cancer Resection. Gastroenterology. 2023 Dec;165(6):1430-1442.e14. doi: 10.1053/j.gastro.2023.08.022. Epub 2023 Aug 23. PMID 37625498